CLINICAL TRIAL: NCT00789750
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Group Study of the Efficacy and Safety of WELCHOL as Add-on to Pioglitazone Therapy for Type 2 Diabetes Mellitus (T2DM)
Brief Title: Colesevelam as Add-on to Pioglitazone Therapy for Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WEL-A-U306
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Colesevelam Hydrochloride; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colesevelam (Experimental): Participants receive six colesevelam tablets (3.8 grams/day) in addition to pioglitazone-based therapy (30 mg or 45 mg)
  Interventions: Drug: Colesevelam; Drug: Pioglitazone
- Placebo (Placebo Comparator): Participants receive six placebo tablets in addition to pioglitazone-based therapy (30 mg or 45 mg)
  Interventions: Drug: Placebo; Drug: Pioglitazone

INTERVENTIONS:
Drug: Colesevelam — Colesevelam 625 mg tablets
  Other Names: Welchol
  Arms: Colesevelam
Drug: Placebo — Placebo tablets appearing to be colesevelam
  Other Names: No drug
  Arms: Placebo
Drug: Pioglitazone — 30 mg or 45 mg pioglitazone therapy
  Other Names: Actos

SUMMARY:
The current study investigates colesevelam as add-on therapy to pioglitazone to improve glycemic control in subjects with type 2 diabetes mellitus not adequately controlled with pioglitazone monotherapy or pioglitazone in combination with either metformin or a sulfonylurea. The study will evaluate if colesevelam add-on to pioglitazone therapy for type 2 diabetes mellitus will be safe, well tolerated, and efficacious.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 diabetes mellitus
* Inadequate glycemic control on a stable dose (at least 2 months prior to screening) of pioglitazone at 30 or 45 mg/day, with or without one or two other oral antidiabetic medications [metformin or a sulfonylurea, or dipeptidyl peptidase (DPP-IV) inhibitor]
* Hemoglobin A1c (HbA1c) >= 7.5% and =< 9.5% at screening
* Fasting plasma glucose =<240 mg/dL at randomization (Week 0/Day 1).
* Male or female >= 18 years of age.
* Women of childbearing potential must be using an adequate method of contraception as detailed per-protocol
* Fasting C-peptide level >0.5 ng/mL at screening
* Clinically stable in regards to medical conditions other than type 2 diabetes
* Concomitant medications are at stable doses for at least 30 days prior to enrollment, and are not anticipated to need adjustment during the study period

Exclusion Criteria:

* History of Type 1 diabetes and/or history of ketoacidosis
* History of bowel obstruction
* History of hypertriglyceridemia-induced pancreatitis
* Fasting serum triglyceride concentration >500 mg/dL
* History of dysphagia, swallowing disorders, gastroparesis, other gastrointestinal motility disorders, major gastrointestinal surgery
* History of insulin use >= 2 weeks duration during the previous 3 months or a total of >2 months insulin therapy at any time prior to screening
* Treatment with bile acid sequestrants, including colesevelam within 3 months prior to screening
* Female subject who is pregnant or breastfeeding
* History of unstable angina, myocardial infarction, cerebrovascular accident, transient ischemic attack, or any revascularization within 6 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2009-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (117):
- United States (117):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Green Valley, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Searcy, Arkansas
  - Buena Park, California
  - Burbank, California
  - Chino, California
  - Garden Grove, California
  - Huntington Park, California
  - La Mirada, California
  - Lincoln, California
  - Lomita, California
  - Los Gatos, California
  - Modesto, California
  - San Diego, California
  - Santa Ana, California
  - Tustin, California
  - Walnut Creek, California
  - Coral Gables, Florida
  - DeLand, Florida
  - Delray Beach, Florida
  - Gulf Breeze, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Ormond Beach, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Sanford, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Wellington, Florida
  - Winter Haven, Florida
  - Winter Park, Florida
  - Columbus, Georgia
  - Decatur, Georgia
  - East Point, Georgia
  - Marietta, Georgia
  - Roswell, Georgia
  - Stockbridge, Georgia
  - Tucker, Georgia
  - Waycross, Georgia
  - Nampa, Idaho
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Bloomington, Indiana
  - Evansville, Indiana
  - La Porte, Indiana
  - South Bend, Indiana
  - Crestview Hills, Kentucky
  - Paducah, Kentucky
  - Lafayette, Louisiana
  - Prince Frederick, Maryland
  - Silver Spring, Maryland
  - New Bedford, Massachusetts
  - Southfield, Michigan
  - Brooklyn Center, Minnesota
  - Jackson, Mississippi
  - Port Gibson, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Las Vegas, Nevada
  - Belvidere, New Jersey
  - Berlin, New Jersey
  - Clifton, New Jersey
  - Lumberton, New Jersey
  - Mine Hill, New Jersey
  - New Windsor, New York
  - North Massapequa, New York
  - Tonawanda, New York
  - West Seneca, New York
  - Lexington, North Carolina
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Cuyahoga Falls, Ohio
  - Marion, Ohio
  - Shaker Heights, Ohio
  - Stow, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Harrisburg, Pennsylvania
  - Jersey Shore, Pennsylvania
  - Philadelphia, Pennsylvania
  - Upper Saint Clair, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greer, South Carolina
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Murfreesboro, Tennessee
  - New Tazewell, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Grand Prairie, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - Alexandria, Virginia
  - Danville, Virginia
  - Manassas, Virginia
  - Richmond, Virginia
  - Salem, Virginia
  - Suffolk, Virginia
  - Lakewood, Washington
  - Kenosha, Wisconsin

REFERENCES:
- [Derived] Rosenstock J, Truitt KE, Baz-Hecht M, Ford DM, Tao B, Chou HS. Efficacy and safety of colesevelam in combination with pioglitazone in patients with type 2 diabetes mellitus. Horm Metab Res. 2014 Dec;46(13):943-9. doi: 10.1055/s-0034-1383648. Epub 2014 Jul 23. PMID 25054436

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The safety set includes all randomized participants who took at least one dose of study medication and have at least one post-baseline safety measurement.
  The intent-to-treat set includes all randomized subjects who took at least one dose of study medication, and had a baseline and at least one post-baseline HbA1c or FPG measurement.
Pre-assignment Details: There was a lead-in period that occurred after participant enrollment, but before randomization.1538 were screened, and a total of 562 participants were randomized.
Groups:
- Colesevelam: Colesevelam tablets with pioglitazone therapy
- Placebo: Placebo tablets with pioglitazone therapy
Period: Overall Study
Arm/Group | Colesevelam | Placebo
Started | 280 | 282
Dropped During run-in Period | 6 | 5
Safety Set | 274 | 277
Intent to Treat Set | 271 | 276
Completed | 221 | 222
Not Completed | 59 | 60

BASELINE CHARACTERISTICS:
Population: All subjects randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Colesevelam | Placebo | Total
Number analyzed (Participants) | 280 | 282 | 562
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 220 | 222 | 442
  >=65 years | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.22) | 55.6 (10.61) | 56.0 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 106 | 242
  Male | 144 | 176 | 320
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 179 | 172 | 351
  Black | 59 | 56 | 115
  Asian | 23 | 30 | 53
  American Indian or Alaskan Native | 16 | 21 | 37
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Other | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 280 | 282 | 562

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 24
Time Frame: Baseline, Week 24
Population: Intent-to-treat, last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 271 | 276
percent | -0.34 (0.083) | -0.02 (0.083)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.49 to -0.16], Standard Error of Mean 0.084

2. Secondary Outcome: Change From Baseline in HbA1c at Week 4
Time Frame: Baseline, Week 4
Population: Intent to treat set, with baseline and post-baseline measures at the given time point
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 264 | 266
percent | -0.28 (0.037) | -0.11 (0.037)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.24 to -0.10], Standard Error of Mean 0.037

3. Secondary Outcome: Change From Baseline in HbA1c at Week 8
Time Frame: Baseline, Week 8
Population: Intent to treat set, with baseline and post-baseline measures at the given time point
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 256 | 256
percent | -0.35 (0.055) | -0.14 (0.056)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.32 to -0.10], Standard Error of Mean 0.056

4. Secondary Outcome: Change From Baseline in HbA1c at Week 16
Time Frame: Baseline, Week 16
Population: Intent to treat set, with baseline and post-baseline measures at the given time point
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 232 | 232
percent | -0.50 (0.078) | -0.15 (0.078)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.51 to -0.20], Standard Error of Mean 0.077

5. Secondary Outcome: Number of Participants Achieving an HbA1c Goal of <7.0%
Time Frame: Week 24
Population: Intent-to-treat set, with last observation carried forward
Measure: Count of Participants; unit: Participants
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 271 | 276
Participants | 56 | 35
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Test type: Other; p = 0.012, Cochran-Mantel-Haenszel

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: In this study a reduction in FPG of at least 30 mg/dL is considered glycemic response.
Time Frame: Baseline, Week 24
Population: Participants in the intent-to-treat set with values at both baseline and Week 24 with last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 268 | 270
mg/dL | -4.8 (3.66) | 9.9 (3.66)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -14.7, 95% CI 2-sided [-21.93 to -7.49], Standard Error of Mean 3.68

7. Secondary Outcome: Number of Participants With a Decrease of >= 0.7 Percent in HbA1c
Time Frame: Week 24
Population: Intent-to-treat set, with last count carried forward
Measure: Count of Participants; unit: Participants
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 271 | 276
Participants | 108 | 70
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Test type: Other; p = 0.0003, Cochran-Mantel-Haenszel

8. Secondary Outcome: Number of Participants With a Decrease of >= 0.5 Percent in HbA1c
Time Frame: Week 24
Population: Intent-to-treat set, with last count carried forward
Measure: Count of Participants; unit: Participants
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 271 | 276
Participants | 147 | 106
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel

9. Secondary Outcome: Number of Participants With a Reduction in FPG of >= 30 mg/dL
Time Frame: Week 24
Population: Intent-to-treat set, with last count carried forward
Measure: Count of Participants; unit: Participants
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 271 | 276
Participants | 60 | 47
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Test type: Other; p = 0.132, Cochran-Mantel-Haenszel

10. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC)
Description: TC is measured in milligrams per deciliter (mg/dL)
Time Frame: Baseline, Week 24
Population: Intent-to-treat set, with values at both baseline and Week 24 with last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 263 | 263
percentage of change | -3.4 (1.33) | 3.1 (1.32)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Test type: Other; p < 0.001, ANCOVA

11. Secondary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: LDL-C is measured in mg/dL
Time Frame: Baseline, Week 24
Population: Intent-to-treat set, with values at both baseline and Week 24 with last count carried forward
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 262 | 263
percentage of change | -9.1 (2.14) | 7.3 (2.12)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -16.4, 95% CI 2-sided [-20.62 to -12.18], Standard Error of Mean 2.15

12. Secondary Outcome: Percent Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C)
Description: HDL-C is measured in mg/dL
Time Frame: Baseline, Week 24
Population: Intent-to-treat set, with values at both baseline and Week 24 with last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 263 | 263
percentage of change | 2.9 (1.30) | 1.1 (1.30)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p = 0.1652, ANCOVA; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-0.75 to 4.39], Standard Error of Mean 1.31

13. Secondary Outcome: Percent Change From Baseline in Non-HDL-C
Description: Non-HDL-C is measured in mg/dL
Time Frame: Baseline, Week 24
Population: Intent-to-treat set, with values at both baseline and Week 24 with last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 263 | 263
percentage of change | -5.2 (1.85) | 4.6 (1.84)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -9.8, 95% CI 2-sided [-13.44 to -6.16], Standard Error of Mean 1.85

14. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG)
Description: TG are measured in mg/dL
Time Frame: Baseline, Week 24
Population: Intent-to-treat set, with values at both baseline and Week 24 with last observation carried forward
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 263 | 263
percentage of change | 14.1 [-4.32 to 32.52] | 2.2 [-14.6 to 19.0]
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p = 0.0004, ANCOVA; Median Difference (Final Values) = 11.3, 95% CI 2-sided [5.3 to 17.5], Standard Error of Mean 67.01 — The treatment difference and its 95% confidence interval are estimated using the Hodges-Lehmann estimator and Moses method. The parameter dispersion Type is actually IQR of the Median Difference

15. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 (Apo A-I)
Description: Apo A-1 is measured in mg/dL
Time Frame: Baseline, Week 24
Population: Intent-to-treat, with values at both baseline and Week 24 with last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 263 | 262
percentage of change | 3.2 (0.92) | -0.2 (0.92)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [1.58 to 5.23], Standard Error of Mean 0.93

16. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B)
Description: Apo B is measured in mg/dL
Time Frame: Baseline, Week 24
Population: Intent-to-treat set, with values at both baseline and Week 24 with last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 263 | 262
percentage of change | -5.2 (1.51) | 3.6 (1.51)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -8.8, 95% CI 2-sided [-11.75 to -5.78], Standard Error of Mean 1.52

17. Secondary Outcome: Change From Baseline in Fasting Insulin Levels
Time Frame: Baseline, Week 24
Population: Intent-to-treat set, with values at both baseline and Week 24 with last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: µIU/mL
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 246 | 248
µIU/mL | 0.2 (1.76) | 0.8 (1.76)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p = 0.7286, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-4.1 to 2.9], Standard Error of Mean 1.77

18. Secondary Outcome: Change From Baseline in Fasting C-peptide
Time Frame: Baseline, Week 24
Population: Intent-to-treat set, with values at both baseline and Week 24 with last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 253 | 255
ng/mL | 0.1 (0.10) | 0.3 (0.10)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p = 0.0653, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.11

19. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: HOMA-IR is a calculation of fasting insulin and fasting glucose that shows the level of insulin resistance. Lower numbers are better.
Time Frame: Baseline, Week 24
Population: Intent-to-treat set, with values at both baseline and Week 24 with last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: calculation
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 227 | 227
calculation | 0.2 (0.71) | 0.3 (0.72)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; Treatment difference = Colesevelam - Placebo; Test type: Other; p = 0.8862, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.5 to 1.3], Standard Error of Mean 0.73

ADVERSE EVENTS:
Time Frame: Adverse events that first occurred or worsened in severity after initiation of treatment with the investigational product and up to the end of study assessment and follow-up period, within 3 years, 3 months
Description: Four potential cardiac events were referred to the Clinical Event Committee (CEC) for adjudication: 1 event was adjudicated as stroke and was considered unrelated to study treatment, while 3 were adjudicated as noncardiac chest pain. No serious adverse events in either treatment group were considered drug-related.
Arm/Group | Colesevelam | Placebo
All-Cause Mortality (participants affected / at risk) | 0/274 | 0/277
Serious Adverse Events (participants affected / at risk) | 11/274 | 4/277
Other Adverse Events (participants affected / at risk) | 11/274 | 17/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Colesevelam (N=274) | Placebo (N=277)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Colesevelam (N=274) | Placebo (N=277)
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees to wait until after coordinated multicenter publication or one year after the trial is over, whichever occurs first. After such time, Study Site will submit any publication to DSI for CCI review and comment at least forty-five (45) days prior to submission. Site agrees to delay publication for an additional sixty (60) days for legal (e.g., patent) concerns. Nothing shall be taken as giving DSI any right of editorial control over any publication prepared by Study Site.